CLINICAL TRIAL: NCT00934167
Title: NON CLINICAL INFERIORITY OF HEPARIN SODIUM PRODUCED BY HIPOLABOR FARMACEUTICA LTDA COMPARED TO THE HEPARIN SODIUM PRODUCED BY APP PHARMACEUTICALS IN VENOUS THROMBOEMBOLISM PROPHYLAXIS, IN SURGICAL PATIENTS WITH MEDIUM RISK FOR DEVELOPMENT OF THROMBOEMBOLISM.
Brief Title: Efficacy of Sodium Heparin for Prophylaxis of Venous Thromboembolism in Surgical Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HEPHIP0509_PRO; Version 01 - AMENDMENT 01; JAN. 2010
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-02

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Hipolabor
  Interventions: Biological: heparin sodium - Hipolabor
- Comparator (Active Comparator): 5.000 USP/mL - APP
  Interventions: Biological: Heparin sodium - APP

INTERVENTIONS:
Biological: heparin sodium - Hipolabor — 5.000 UI/0,25mL
  Arms: Test
Biological: Heparin sodium - APP — 5.000 USP/mL
  Arms: Comparator

SUMMARY:
The aim of this study is to verify, through clinical examination and doppler, the non-inferiority of the drug test (heparin sodium 5.000UI/0.25 mL - HIPOLABOR) in relation to the drug compared (heparin sodium 5.000USP/mL - APP) in preventing the development of venous thromboembolism (VTE) in patients undergoing surgery for medium risk for the development of this pathology.

ELIGIBILITY:
Inclusion Criteria:

* Accept all items described in IC signing it in two ways;
* Be aged between 18 and 60;
* Be alert to the need for surgery antithrombotic prophylaxis;
* Be classified as "moderate risk" for developing VTE, according to the protocol of prophylaxis of deep vein thrombosis of the Brazilian Society of Angiology and Vascular Surgery.

Exclusion Criteria:

* Acute coronary syndrome, it will make use of anticoagulation;
* Immobilization of the lower limbs due to fractures, because in this way will be considered as high risk;
* History of recent stroke;
* Patients at high risk of bleeding in which the use of heparin is contra-indicated;
* General Surgery in patients over 60 years in the case of patients at high risk for VTE;
* general surgery in patients 40 to 60 years with additional risk factors for development of VTE;
* Major amputations;
* More orthopedic surgeries;
* Patients with pre-surgical diagnosis of malignant neoplasms;
* Patients with a platelet level below 100x109 / L;
* Use of anticoagulants 48 hours before randomization;
* Severe liver failure;
* Be classified as "Low Risk" or "high risk" for developing VTE, according to Maffei et al. (2005);
* Pregnancy and lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-11 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Non-appearance of venous thromboembolism | 2 h before the start of surgery, 1, 2, 3, 4, 5, 6, 7, 14, 21, 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Lal Clinica Pesquisa E Desenvolvimento Ltda, Valinhos, São Paulo, Brazil